CLINICAL TRIAL: NCT01380717
Title: The Role of Renal and Peripheral Vascular Resistance in Chronic Kidney Disease
Brief Title: Renal and Systemic Vascular Resistance in Chronic Kidney Disease (CKD)
Acronym: RenVas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenVas
Record Dates: First submitted 2011-06-20; First posted 2011-06-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Kidney Insufficiency; Hypertension; Vasodilation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Aneurysm | interventions — Adrenergic beta-Antagonists; Angiotensin-Converting Enzyme Inhibitors; Calcium Channel Blockers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment (Active Comparator): Patients with CKD 3-4, hypertension, treated for 18 months with beta-blocker and if needed ACE-inhibitor or ARB.
  Interventions: Drug: Beta-blocker, ACE-inhibitor
- Intensive vasodilation (Active Comparator): Patients with CKD 3-4 and hypertension, randomized to treatment with calcium channel blocker and if needed ACE-inhibitor or ARB for 18 months
  Interventions: Drug: Calcium Channel Blockers, ACE-Inhibitor

INTERVENTIONS:
Drug: Beta-blocker, ACE-inhibitor — Beta-blocker: 50- 100 mg 1-2 times a day. ACEi: 5-10 mg once a day
  Arms: Standard treatment
Drug: Calcium Channel Blockers, ACE-Inhibitor — Calcium Channel Blockers: 5-10 mg a day. ACEi: 5-10 mg a day
  Arms: Intensive vasodilation

SUMMARY:
Patients with reduced kidney function have a higher risk of heart disease and death. Studies have shown that blood vessels in patients with hypertension change with a decrease of lumen size and growth of the vessel wall. By treating patients with antihypertensive certain medication vessel lumen and walls normalize. Treating hypertension in patients with chronic kidney disease slows the progression of kidney function loss.

The aim is to compare different degrees of antihypertensive medication in patients with chronic kidney disease and hypertension will slow the progression of kidney loss.

ELIGIBILITY:
Inclusion Criteria:

* eGFR 15-60 ml/min for at least 3 months
* Blood pressure > 130 mmHg systolic og >80 mmHg diastolic (patients without antihypertensive treatment or in treatment with Beta-blockers, ACEi, ARBs or CCB not in maximum dosi).
* Blood pressure < 130 mmHg systolic og < 80 mmHg diastolic (patients receiving Beta-blockers, ACEi, ARBs og CCB).
* Fertile women using safe contraceptives

Exclusion Criteria:

* Ultrasound verified Polycystic Kidney Disease (ADPKD)
* Claustrophobia (MRi scan).
* Contraindications to MRi.
* Pregnancy or wish to become pregnant in the study period.
* Nephrotic syndrome with gross edema.
* Known allergy to any study medication.
* Blood pressure < 130 mmHg systolic or < 80 mmHg diastolic without antihypertensive treatment.
* Blood pressure > 130 mmHg systolic or > 80 mmHg diastolic and in maximum dosages of all three Beta-blockers, ACEi (ARBs) and CCB.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in glomerular filtration rate between the two treatment arms. | Measured at baseline and after 18 months of treatment

SECONDARY OUTCOMES:
Changes in glomerular filtration rate stratified after changes in pulse wave velocity, renal vascular resistance and forearm minimal resistance at baseline and after 18 months of treatment. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Niels Henrik Buus, DrMedSc, Principal Investigator — Department og Renal Medicine, Aarhus University Hospital, Skejby
Locations (1):
- Department of Renal Medicine, Aarhus University Hospital, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Svendsen SL, Rousing AQ, Carlsen RK, Khatir D, Jensen D, Hansen NM, Salomo L, Birn H, Buus NH, Leipziger J, Sorensen MV, Berg P. A Urine pH-Ammonium Acid/Base Score and CKD Progression. J Am Soc Nephrol. 2024 Nov 1;35(11):1533-1545. doi: 10.1681/ASN.0000000000000447. Epub 2024 Jul 17. PMID 39485702